**Study:** A Feasibility Study of Integrating Maternal Nutrition Interventions into Antenatal Care Services in Ethiopia: A Cluster-Randomized Evaluation

Clinicaltrials.gov: NCT04155437

Document date: November 16, 2020

**PHASE:** Endline survey

### INFORMATION SHEET (NURSE-MIDWIFE TO OBSERVE THE ANTENATAL CARE SESSION)

Thank you for speaking with us today.

This interview will be held in accordance with COVID-19 prevention measures.

My name is [NAME OF INTERVIEWER]. I am a member of a survey team from Agence de Formation, de Recherche & d'Expertise en Santé (AFRICSanté), a research organization in Bobo-Dioulasso. Together with the International Food Policy Research Institute (IFPRI), we are studying the Alive & Thrive program on maternal nutrition in this area. Your facility was selected to participate in this study.

A baseline survey was conducted in November and December 2019 for CSPSs and households. At the household level, 960 pregnant women and 1920 mothers of children 0-5 months old were interviewed. At CSPS level, antenatal care (ANC) consultations of 160 pregnant women were observed and the women were interviewed. Pregnant women were asked about the messages they received and their level of satisfaction with the care received. When the baseline survey was completed, maternal nutrition interventions were implemented in some health centers and villages for 12 months. The final survey that we are about to start will consist of collecting similar information to assess the impact of these interventions on pregnant women and mothers of children 0-5 months.

We will be observing two ANC consultations today. Information collected during this observation will be used to improve maternal nutrition through antenatal care services in this community and across Burkina Faso. Your participation is voluntary.

During the prenatal consultations, we will be present in the room only to observe. You can do the prenatal consultation as normal, without worrying about our presence. We will ask for the consent of the pregnant woman before the start of each consultation. You and the pregnant woman can ask us to stop observing at any time during the consultation. Your decision to participate or not will not affect your work at the CSPS. For her time spent answering our questions at the end of the consultation, we will give the pregnant woman 500 CFA francs as compensation.

Do not worry about telling us your name, because we will not keep it. We are asking for it only to get to know you before the conversation. You will not be identified by your name. With your permission, we will take notes during the observation and no one will have access to the notes of our observations except the research team.

Contact with our survey team presents a risk of spreading COVID-19, an illness that can spread from person to person. To protect you, our survey team members will maintain two meters of distance, wear a mask, and wash or sanitize hands before and after the interview. We will also provide you with a mask. Each member of our survey team was checked for any symptoms of COVID-19 before starting work today. We ask that you let us know whether you have experienced any COVID-19 related symptoms today, so that additional safety measures can be applied if needed.

If you have any questions concerning the study, you may ask questions at any time before agreeing to participate or during the observation, or you can talk with:

Dr. Rasmané Ganaba Director AFRICSanté 01 BP 298 Bobo-Dioulasso Phone: +226 20 986 368 | Email: rganaba@hotmail.com

Dr. Lieven Huybregts Research Fellow and IRB Chair International Food Policy Research Institute

Address: 1201 Eye St. NW, Washington, DC 20005-3915 USA

Tel: +1 202-862-6481 | Email: <u>I.huybregts@cgiar.org</u>

The Chairmen of the ethics committees which have given their approval:

For the Centre Muraz ethics committee:

Dr. Adama Dembélé: 70 13 68 88

For the IRSS/DRO institutional ethics committee:

## CONSENT OF NURSE-MIDWIFE TO OBSERVE THE ANTENATAL CARE SESSION

The interviewer read to me orally and explained the consent form. I understand that I am free to discontinue participation at any time if I so choose, and that the investigator will gladly answer any questions that arise.

| | Do you agree to participate in this study? | No<br>Yes | | 0<br>1 | | |
|---|---|---|---|---|---|---|
| Nurse | -Midwife's signature: | Date: _ | DAY | MONTH | _/_ | YEAR |
| Interv | iewer's signature: | Date: _ | DAY | / | _/_ | VEAD |

**PHASE:** Endline survey

# INFORMATION SHEET (PREGNANT WOMAN TO PARTICIPATE IN THE ANTENATAL CARE OBSERVATION AND EXIT INTERVIEW)

Thank you for speaking with us today.

This interview will be held in accordance with COVID-19 prevention measures.

My name is [NAME OF INTERVIEWER]. I am a member of a survey team from Agence de Formation, de Recherche & d'Expertise en Santé (AFRICSanté), a research organization in Bobo-Dioulasso. Together with the International Food Policy Research Institute (IFPRI), we are studying the Alive & Thrive program on maternal nutrition in this area.

A baseline survey was conducted in November and December 2019 for CSPSs and households. At the household level, 960 pregnant women and 1920 mothers of children 0-5 months old were interviewed. At CSPS level, antenatal care (ANC) consultations of 160 pregnant women were observed and the women were interviewed. Pregnant women were asked about the messages they received and their level of satisfaction with the care received. When the baseline survey was completed, maternal nutrition interventions were implemented in some health centers and villages for 12 months. The final survey that we are about to start will consist of collecting similar information to assess the impact of these interventions on pregnant women and mothers of children 0-5 months.

We came to you today because you are visiting a CSPS in this area. Your participation is voluntary. Our work today will be conducted in two stages: First, we would like to observe the prenatal consultation you receive. Then, at the end, we would like to ask you some questions.

During the prenatal consultation, we will be present in the room only to observe. You can do the prenatal consultation as normal, without worrying about our presence. The health care provider and you can ask us to stop observing at any time during the consultation. The same is true for the interview that we will conduct with you. You do not have to respond to questions to which you do not wish to respond. You can decide to stop the interview at any time. Your decision to either participate or not will not affect the services and treatments that you receive at the CSPS. For your time spent answering our questions, we will give you 500 CFA francs as compensation.

Do not worry about telling us your name, because we will not keep it. We are asking for it only to get to know you before the conversation. You will not be identified by your name. With your permission, we will take notes during the observation and the interview. No one will have access to the notes of our observations and your responses except the research team.

Contact with our survey team presents a risk of spreading COVID-19, an illness that can spread from person to person. To protect you, our survey team members will maintain two meters of distance, wear a mask, and wash or sanitize hands before and after the interview. We will also provide you with a mask. Each member of our survey team was checked for any symptoms of COVID-19 before starting work today. We ask that you let us know whether you have experienced any COVID-19 related symptoms today, so that additional safety measures can be applied if needed.

If you have any questions concerning the study, you may ask questions at any time before agreeing to participate or during the observation and interview, or you can talk with:

Dr. Rasmané Ganaba

Director AFRICSanté 01 BP 298 Bobo-Dioulasso

Phone: +226 20 986 368 | Email: <u>rganaba@hotmail.com</u>

Dr. Lieven Huybregts
Research Fellow and IRB Chair
International Food Policy Research Institute
Address: 1201 Eye St. NW, Washington, DC 20005-3915 USA
Tel: +1 202-862-6481 | Email: <a href="mailto:l.huybregts@cgiar.org">l.huybregts@cgiar.org</a>

The Chairmen of the ethics committees which have given their approval:

For the ethics committee of Centre Muraz:

Dr. Adama Dembélé: 70 13 68 88

For the IRSS/DRO institutional ethics committee:

# CONSENT FOR PREGNANT WOMAN TO PARTICIPATE IN THE ANTENATAL CARE OBSERVATION AND EXIT INTERVIEW

Use this consent form for all women 18 years of age or older and all married women. If the pregnant woman is not married and is less than 18 years of age, one of her parents/guardians must give consent.

The interviewer read to me orally and explained the consent form. I understand that I am free to discontinue participation at any time if I so choose, and that the investigator will gladly answer any questions that arise.

| | Do you agree to participate in this study? | No<br>Yes | | | | |
|---|---|---|---|---|---|---|
| Pregn | ant woman's signature: | Date | e: | _/_<br>MONTH | | YEAR |
| | t/Guardian's signature:<br>woman is not married and less than 18) | Date | : | /MONTH | _/. | YEAR |
| (if the | ss's signature:<br>woman cannot read or write, an independent w<br>entified and will provide their signature or finger | vitness will | : | _/MONTH | | YEAR |
| Intervi | ewer's signature: | Date: | | /MONTH | _/_ | YEAR |

**PHASE:** Endline survey

#### **INFORMATION SHEET (COMMUNITY HEALTH WORKER)**

Thank you for speaking with us today.

This interview will be held in accordance with COVID-19 prevention measures.

My name is [NAME OF INTERVIEWER]. I am a member of a survey team from the Agence de Formation, de Recherche & d'Expertise en Santé (AFRICSanté), a research organization based in Bobo-Dioulasso. Together with the International Food Policy Research Institute (IFPRI), we are studying the Alive & Thrive program on maternal nutrition in this area.

We want to talk with you about the services that you provide at this CSPS and your community. We will also be asking you questions about training and supervision that you received. The information that you provide us will be used to improve maternal nutrition through antenatal care services in this area and across Burkina Faso.

A baseline survey was conducted in November and December 2019 for CSPSs and households. At the household level, 240 community health workers (ASBCs) were interviewed. ASBCs were asked about their workload, knowledge of maternal and child health and nutrition, training, and supervision. When the baseline survey was completed, maternal nutrition interventions were implemented in some health centers and villages for 12 months. The final survey that we are about to start will consist of collecting similar information to assess the impact of these interventions on pregnant women and mothers of children 0-5 months.

The interview may last for about one hour. The information you will give us will not be disclosed to anyone. It will be kept strictly confidential.

Your participation in the interview is voluntary. You have the right not to participate if you do not want to. You also have the right to decline to answer specific questions or to stop this interview at any point during the interview. Not participating will not affect you or your work. For your time spent answering our questions, we will give you 1000 CFA francs as compensation.

Contact with our survey team presents a risk of spreading COVID-19, an illness that can spread from person to person. To protect you, our survey team members will maintain two meters of distance, wear a mask, and wash or sanitize hands before and after the interview. We will also provide you with a mask. Each member of our survey team was checked for any symptoms of COVID-19 before starting work today. We ask that you let us know whether you have experienced any COVID-19 related symptoms today, so that additional safety measures can be applied if needed.

Your participation will be highly appreciated. The answers you give will help provide better information to policymakers and practitioners so that they can plan for better services that will respond to your needs.

If you have any questions concerning the study, you may ask questions at any time before agreeing to participate or during the interview, or you can talk with:

Dr. Rasmané Ganaba Director AFRICSanté 01 BP 298 Bobo-Dioulasso

Phone: +226 20 986 368 | Email: <u>rganaba@hotmail.com</u>

Dr. Lieven Huybregts Research Fellow and IRB Chair International Food Policy Research Institute Address: 1201 Eye St. NW, Washington, DC 20005-3915 USA

Tel: +1 202-862-6481 | Email: <u>l.huybregts@cgiar.org</u>

The Chairmen of the ethics committees which have given their approval:

For the Centre Muraz ethics committee:

Dr. Adama Dembélé: 70 13 68 88

For the IRSS/DRO institutional ethics committee:

# CONSENT OF RESPONDENT (COMMUNITY HEALTH WORKER)

The interviewer read to me orally and explained the consent form. I understand that I am free to discontinue participation at any time if I so choose, and that the investigator will gladly answer any questions that arise.

| Do you agree to participate in this study? | No<br>Yes | | |
|---|---|---|---|
| ASBC's signature: | Date:<br>DA <sup>v</sup> | //// | ₹ |
| Interviewer's signature: | Date: | ///////// | |

**PHASE:** Endline survey

### **INFORMATION SHEET (HUSBAND)**

Thank you for speaking with us today.

This interview will be held in accordance with COVID-19 prevention measures.

My name is [NAME OF INTERVIEWER]. I am a member of a survey team from Agence de Formation, de Recherche & d'Expertise en Santé (AFRICSanté), a research organization based in Bobo-Dioulasso. Together with the International Food Policy Research Institute (IFPRI), we are studying the Alive & Thrive program on maternal nutrition in this area.

We want to talk with you about health and nutrition during pregnancy. We will also be asking you questions about your household. The information that you provide us will be used to improve maternal nutrition through antenatal care services in this community and across Burkina Faso.

A baseline survey was conducted in November and December 2019 for CSPSs and households. At the household level, 960 pregnant women and 1920 mothers of children 0-5 months old and their husbands were interviewed. Husbands were asked about their support during pregnancy, exposure to maternal nutrition information, and their knowledge and perceptions of maternal nutrition. When the baseline survey was completed, maternal nutrition interventions were implemented in some health centers and villages for 12 months. The final survey that we are about to start will consist of collecting similar information to assess the impact of these interventions on pregnant women and mothers of children 0-5 months.

The interview may last for one hour. The information you will give us will not be disclosed to anyone. It will be kept strictly confidential. No matter how you answer our questions, you and your family will continue to receive all services that you normally receive through health facilities and from community health workers.

Your participation in the interview is voluntary. You have the right to not participate if you do not want to. You also have the right to refuse to answer specific questions or to stop this interview at any point during the interview. Not participating will not affect you or your family. For your time spent answering our questions, we will give you 1000 CFA francs as compensation.

Contact with our survey team presents a risk of spreading COVID-19, an illness that can spread from person to person. To protect you, our survey team members will maintain two meters of distance, wear a mask, and wash or sanitize hands before and after the interview. We will also provide you with a mask. Each member of our survey team was checked for any symptoms of COVID-19 before starting work today. We ask that you let us know whether you have experienced any COVID-19 related symptoms today, so that additional safety measures can be applied if needed.

Your participation will be highly appreciated. The answers you give will help provide better information to policymakers and practitioners so that they can plan for better services that will respond to your needs.

If you have any questions concerning the study, you may ask questions at any time before agreeing to participate or during the interview, or you can talk with:

Dr. Rasmané Ganaba Director AFRICSanté 01 BP 298 Bobo-Dioulasso

Phone: +226 20 986 368 | Email: <u>rganaba@hotmail.com</u>

Dr. Lieven Huybregts Research Fellow and IRB Chair International Food Policy Research Institute

Address: 1201 Eye St. NW, Washington, DC 20005-3915 USA

Tel: +1 202-862-6481 | Email: <u>l.huybregts@cgiar.org</u>

The Chairmen of the ethics committees which have given their approval:

For the Centre Muraz ethics committee:

Dr. Adama Dembélé: 70 13 68 88

For the IRSS/DRO institutional ethics committee:

## **CONSENT OF RESPONDENT (HUSBAND)**

| Member ID (from 201) |
|----------------------|
|----------------------|

The researcher read to me orally and explained the consent form. I understand that I am free to discontinue participation at any time if I so choose, and that the investigator will gladly answer any questions that arise.

| | Do you agree to participate in this study? No | | | | |
|---|---|---|---|---|---|
| Husba | nd's signature: | Date: _ | DAY | _//<br>/ | YEAR |
| Intervi | ewer's signature: | Date: | | 1 1 | |
| | | | DAY | MONTH | YEAR |

**PHASE:** Endline survey

#### **INFORMATION SHEET (HEAD OF CSPS)**

Thank you for speaking with us today.

This interview will be held in accordance with COVID-19 prevention measures.

My name is [NAME OF INTERVIEWER]. I am a member of a survey team from the Agence de Formation, de Recherche & d'Expertise en Santé (AFRICSanté), a research organization based in Bobo-Dioulasso. Together with the International Food Policy Research Institute (IFPRI), we are studying the Alive & Thrive program on maternal nutrition in this area.

A baseline survey was conducted in November and December 2019 for CSPSs and households. At the CSPS level, 80 CSPS were included. Information was collected on the infrastructure, characteristics of facilities and personnel, equipment, materials and drugs used for providing ANC, ANC services provided, staff workloads, and ANC monitoring systems. When the baseline survey was completed, maternal nutrition interventions were implemented in some health centers and villages for 12 months. The final survey that we are about to start will consist of collecting similar information to assess the impact of these interventions.

Your facility was selected to participate in this study. We will be making some observations of the CSPS and will ask you questions about health services provided at this facility. Information collected about your facility during this study will be used to improve maternal nutrition through antenatal care services in this community and across Burkina Faso.

The observation will last for about one hour. The information you will give us will not be disclosed to anyone. It will be kept strictly confidential.

Your participation in the interview is voluntary. You may refuse to answer any question or choose to stop the interview at any time. Not participating will not affect you or your work. For your time spent answering our questions, we will give you 1000 CFA francs as compensation.

Contact with our survey team presents a risk of spreading COVID-19, an illness that can spread from person to person. To protect you, our survey team members will maintain two meters of distance, wear a mask, and wash or sanitize hands before and after the interview. We will also provide you with a mask. Each member of our survey team was checked for any symptoms of COVID-19 before starting work today. We ask that you let us know whether you have experienced any COVID-19 related symptoms today, so that additional safety measures can be applied if needed.

Your participation will be highly appreciated. The answers you give will help provide better information to policymakers and practitioners so that they can plan for better services that will respond to your needs.

If there are questions for which someone else is the most appropriate person to provide the information, we would appreciate it if you introduce us to that person to help us collect that information.

If you have any questions concerning the study, you may ask questions at any time before agreeing to participate or during the interview, or you can talk with:

Dr. Rasmané Ganaba Director AFRICSanté 01 BP 298 Bobo-Dioulasso

Phone: +226 20 986 368 | Email: <u>rganaba@hotmail.com</u>

Dr. Lieven Huybregts Research Fellow and IRB Chair International Food Policy Research Institute

Address: 1201 Eye St. NW, Washington, DC 20005-3915 USA

Tel: +1 202-862-6481 | Email: <u>l.huybregts@cgiar.org</u>

The Chairmen of the ethics committees which have given their approval:

For the Centre Muraz ethics committee:

Dr. Adama Dembélé: 70 13 68 88

For the IRSS/DRO institutional ethics committee:

## **CONSENT OF RESPONDENT (HEAD OF CSPS)**

The interviewer read to me orally and explained the consent form. I understand that I am free to discontinue participation at any time if I so choose, and that the interviewer will gladly answer any questions that arise.

| | Do you agree to participate in this study? | No<br>Yes | | | | |
|---|---|---|---|---|---|---|
| Respo | ndent's signature: | Date: | <br>DAY | / | ./_ | YEAR |
| Intervi | ewer's signature: | Date: | DAY | / | _/ | YΕΔR |

**PHASE:** Endline survey

## **INFORMATION SHEET (NURSE-MIDWIFE)**

Thank you for speaking with us today.

This interview will be held in accordance with COVID-19 prevention measures.

My name is [NAME OF INTERVIEWER]. I am a member of a survey team from the Agence de Formation, de Recherche & d'Expertise en Santé (AFRICSanté), a research organization based in Bobo-Dioulasso. Together with the International Food Policy Research Institute (IFPRI), we are studying the Alive & Thrive program on maternal nutrition in this area.

We want to talk with you about the services that you provide at this CSPS. We will also be asking you questions about training and supervision that you received. The information that you provide us will be used to improve maternal nutrition through antenatal care services in this area and across Burkina Faso.

A baseline survey was conducted in November and December 2019 for CSPSs and households. At the CSPS level, 80 nurse-midwives were interviewed. Nurse-midwives were asked about their workload, knowledge of maternal and child health and nutrition, training, and supervision. When the baseline survey was completed, maternal nutrition interventions were implemented in some health centers and villages for 12 months. The final survey that we are about to start will consist of collecting similar information to assess the impact of these interventions.

The interview may last for about one hour. The information you will give us will not be disclosed to anyone. It will be kept strictly confidential.

Your participation in the interview is voluntary. You have the right to not participate if you do not want to. You also have the right to refuse to answer specific questions or to stop this interview at any point during the interview. Not participating will not affect you or your work. For your time spent answering our questions, we will give you 1000 CFA francs as compensation.

Contact with our survey team presents a risk of spreading COVID-19, an illness that can spread from person to person. To protect you, our survey team members will maintain two meters of distance, wear a mask, and wash or sanitize hands before and after the interview. We will also provide you with a mask. Each member of our survey team was checked for any symptoms of COVID-19 before starting work today. We ask that you let us know whether you have experienced any COVID-19 related symptoms today, so that additional safety measures can be applied if needed.

Your participation will be highly appreciated. The answers you give will help provide better information to policymakers and practitioners so that they can plan for better services that will respond to your needs.

If you have any questions concerning the study, you may ask questions at any time before agreeing to participate or during the interview, or you can talk with:

Dr. Rasmané Ganaba Director AFRICSanté 01 BP 298 Bobo-Dioulasso

Phone: +226 20 986 368 | Email: rganaba@hotmail.com

Dr. Lieven Huybregts

Research Fellow and IRB Chair International Food Policy Research Institute

Address: 1201 Eye St. NW, Washington, DC 20005-3915 USA

Tel: +1 202-862-6481 | Email: <a href="mailto:l.huybregts@cgiar.org">l.huybregts@cgiar.org</a>

The Chairmen of the ethics committees which have given their approval:

For the Centre Muraz ethics committee:

Dr. Adama Dembélé: 70 13 68 88

For the IRSS/DRO institutional ethics committee:

# CONSENT OF RESPONDENT (NURSE-MIDWIFE)

The interviewer read to me orally and explained the consent form. I understand that I am free to discontinue participation at any time if I so choose, and that the interviewer will gladly answer any questions that arise.

| Do you agree to participate in this study? | No 0<br>Yes 1 | |
|--------------------------------------------|-------------------|------|
| Nurse-Midwife's signature: | / Date://// | YEAR |
| Interviewer's signature: | Date: / / / / / / | VΕΔR |

**PHASE:** Endline survey

#### **INFORMATION SHEET (PREGNANT WOMAN)**

Thank you for speaking with us today.

This interview will be held in accordance with COVID-19 prevention measures.

My name is [NAME OF INTERVIEWER]. I am a member of a survey team from Agence de Formation, de Recherche & d'Expertiseen Santé (AFRICSanté), a research organization based in Bobo-Dioulasso. Together with the International Food Policy Research Institute (IFPRI), we are studying the Alive & Thrive program on maternal nutrition in this area.

We want to talk with you about your health and nutrition during pregnancy. We will also be asking you questions about your household. The information that you provide us will be used to improve maternal nutrition through antenatal care services in this community and across Burkina Faso.

A baseline survey was conducted in November and December 2019 for CSPSs and households. At the household level, 960 pregnant women and 1920 mothers of children 0-5 months old were interviewed. Pregnant women and mothers were asked about household composition, socioeconomic status, food security, obstetrical history, use of and exposure to antenatal care, maternal nutrition and breastfeeding knowledge, desire for social acceptance, decision-making power, and mental health. When the baseline survey was completed, maternal nutrition interventions were implemented in some health centers and villages for 12 months. The final survey that we are about to start will consist of collecting similar information to assess the impact of these interventions on pregnant women and mothers of children 0-5 months.

The interview may last for about two hours. The information you will give us will not be disclosed to anyone. It will be kept strictly confidential. No matter how you answer our questions, you will continue to receive all services that you normally receive through health facilities and from community health workers.

Your participation in the interview is voluntary. You have the right to not participate if you do not want to. You also have the right to refuse to answer specific questions or to stop this interview at any point during the interview. Not participating will not affect you or your family. For your time spent answering our questions, we will give you 1000 CFA francs as compensation.

Contact with our survey team presents a risk of spreading COVID-19, an illness that can spread from person to person. To protect you, our survey team members will maintain two meters of distance, wear a mask, and wash or sanitize hands before and after the interview. We will also provide you with a mask. Each member of our survey team was checked for any symptoms of COVID-19 before starting work today. We ask that you let us know whether you have experienced any COVID-19 related symptoms today, so that additional safety measures can be applied if needed.

Your participation will be highly appreciated. The answers you give will help provide better information to policymakers and practitioners so that they can plan for better services that will respond to your needs.

If you have any questions concerning the study, you may ask questions at any time before agreeing to participate or during the interview, or you can talk with:

Dr. Rasmané Ganaba Director AFRICSanté 01 BP 298 Bobo-Dioulasso

Phone: +226 20 986 368 | Email: <u>rganaba@hotmail.com</u>

Dr. Lieven Huybregts Research Fellow and IRB Chair International Food Policy Research Institute

Address: 1201 Eye St. NW, Washington, DC 20005-3915 USA

Tel: +1 202-862-6481 | Email: <u>l.huybregts@cgiar.org</u>

The Chairmen of the ethics committees which have given their approval:

For the ethics committee of Centre Muraz:

Dr. Adama Dembélé: 70 13 68 88

For the IRSS/DRO institutional ethics committee:

## **CONSENT OF RESPONDENT (PREGNANT WOMAN)**

Use this consent form for all women 18 years of age or older and all married women. If the pregnant woman is not married and is less than 18 years of age, one of her parents/guardians must give consent.

The interviewer read to me orally and explained the consent form. I understand that I am free to discontinue participation at any time if I so choose, and that the investigator will gladly answer any questions that arise.

| | Do you agree to participate in this study? | No<br>Yes | | 0 | |
|---|---|---|---|---|---|
| Pregn | ant woman's signature: | Date | E | / MONTH | /YEAR |
| | t/Guardian's signature:<br>woman is not married and less than 18) | Date: | DAY | / | /YEAR |
| (if the | ss's signature:<br>woman cannot read or write, an independent<br>entified and will provide their signature or finge | witness will | : | MONTH | /YEAR |
| Intervi | iewer's signature: | Date: | | //<br>MONTH | /YEAR |

**PHASE:** Endline survey

## INFORMATION SHEET (RECENTLY DELIVERED WOMAN)

Thank you for speaking with us today.

This interview will be held in accordance with COVID-19 prevention measures.

My name is [NAME OF INTERVIEWER]. I am a member of a survey team from Agence de Formation, de Recherche & d'Expertise en Santé (AFRICSanté), a research organization based in Bobo-Dioulasso. Together with the International Food Policy Research Institute (IFPRI), we are studying the Alive & Thrive program on maternal nutrition in this area.

We want to talk with you about health services your received during pregnancy and about health and nutrition during pregnancy. We will also be asking you questions about your household. The information that you provide us will be used to improve maternal nutrition through antenatal care services in this community and across Burkina Faso.

A baseline survey was conducted in November and December 2019 for CSPSs and households. At the household level, 960 pregnant women and 1920 mothers of children 0-5 months old were interviewed. Pregnant women and mothers were asked about household composition, socioeconomic status, food security, obstetrical history, use of and exposure to antenatal care, maternal nutrition and breastfeeding knowledge, desire for social acceptance, decision-making power, and mental health. When the baseline survey was completed, maternal nutrition interventions were implemented in some health centers and villages for 12 months. The final survey that we are about to start will consist of collecting similar information to assess the impact of these interventions on pregnant women and mothers of children 0-5 months.

The interview may last for about two hours. The information you will give us will not be disclosed to anyone. It will be kept strictly confidential. No matter how you answer our questions, you will continue to receive all services that you normally receive through health facilities and from community health workers.

Your participation in the interview is voluntary. You have the right to not participate if you do not want to. You also have the right to refuse to answer specific questions or to stop this interview at any point during the interview. Not participating will not affect you or your family. For your time spent answering our questions, we will give you 1000 CFA francs as compensation.

Contact with our survey team presents a risk of spreading COVID-19, an illness that can spread from person to person. To protect you, our survey team members will maintain two meters of distance, wear a mask, and wash or sanitize hands before and after the interview. We will also provide you with a mask. When conducting height and weight measurements, we will use additional protective equipment, including disposable gloves and overalls. Measuring boards will also be sanitized after every measurement. If you do not want to participate in having your measurements taken, this will not disqualify you from participating in the interview. Each member of our survey team was checked for any symptoms of COVID-19 before starting work today. We ask that you let us know whether you have experienced any COVID-19 related symptoms today, so that additional safety measures can be applied if needed.

Your participation will be highly appreciated. The answers you give will help provide better information to policymakers and practitioners so that they can plan for better services that will respond to your needs.

If you have any questions concerning the study, you may ask questions at any time before agreeing to participate or during the interview, or you can talk with:

Dr. Rasmané Ganaba Director AFRICSanté 01 BP 298 Bobo-Dioulasso

Phone: +226 20 986 368 | Email: <u>rganaba@hotmail.com</u>

Dr. Lieven Huybregts Research Fellow and IRB Chair International Food Policy Research Institute Address: 1201 Eye St. NW, Washington, DC 20005-3915 USA

Tel: +1 202-862-6481 | Email: <a href="mailto:l.huybregts@cgiar.org">l.huybregts@cgiar.org</a>

The Chairmen of the ethics committees which have given their approval:

For the ethics committee of Centre Muraz:

Dr. Adama Dembélé: 70 13 68 88

For the IRSS/DRO institutional ethics committee:

## CONSENT OF RESPONDENT (RECENTLY DELIVERED WOMAN)

Use this consent form for all women 18 years of age or older and all married women. If the recently delivered woman is not married and is less than 18 years of age, one of her parents/guardians must give consent.

The researcher read to me orally and explained the consent form. I understand that I am free to discontinue participation at any time if I so choose, and that the investigator will gladly answer any questions that arise.

| | Do you agree to participate in this study? | No<br>Yes | | _ | |
|---|---|---|---|---|---|
| Recer | ntly delivered woman's signature: | Date: | DAY | //<br> | YEAR |
| | t/Guardian's signature:<br>woman is not married and less than 18) | Date: | DAY | //<br>MONTH | YEAR |
| (if the | ss's signature:<br>woman cannot read or write, an independent<br>entified and will provide their signature or finge | witness will | DAY | / | /YEAR |
| Intervi | ewer's signature: | Date: _ | /<br>DAY | /<br>/ | YEAR |